CLINICAL TRIAL: NCT02624544
Title: Proton Pump Inhibitors Use in Patients With Psoriasis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMS
Record Dates: First submitted 2015-11-13; First posted 2015-12-08 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Esomeprazole; Desonide; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Proton Pump Inhibitor esomeprazole 40 mg twice a day
  Interventions: Drug: esomeprazole
- Group B (Active Comparator): desonide
  Interventions: Drug: desonide

INTERVENTIONS:
Drug: esomeprazole — esomex 40 mg twice daily
  Other Names: esomex
  Arms: Group A
Drug: desonide — topical corticosteroid desonid 0,1% b.i.d
  Other Names: corticosteroid
  Arms: Group B

SUMMARY:
Proton pump inhibitors act in blocking acid secretion and also have antioxidant and anti-inflammatory properties. For that mechanisms possibly PPIs may have an anti-inflammatory action with improvement in skin lesions in patients with psoriasis.

DETAILED DESCRIPTION:
Proton pump inhibitors act in blocking acid secretion and also have antioxidant and anti-inflammatory properties. For that mechanisms possibly PPIs may have an anti-inflammatory action with improvement in skin lesions in patients with psoriasis.

The study will assess the evolution of skin lesions in psoriasis patients using PPIs

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of Psoriasis

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-01 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy - Change from baseline in skin lesions at 5 months | Baseline - 5 months
  Number of Participants With Treatment-Related Clinical Improvement of lesions Change From Baseline in skin lesions at 5 months

REFERENCES:
- [Result] Rahman M, Alam K, Ahmad MZ, Gupta G, Afzal M, Akhter S, Kazmi I, Jyoti, Ahmad FJ, Anwar F. Classical to current approach for treatment of psoriasis: a review. Endocr Metab Immune Disord Drug Targets. 2012 Sep;12(3):287-302. doi: 10.2174/187153012802002901. PMID 22463723